CLINICAL TRIAL: NCT00716703
Title: CT Scan Using IV Contrast Alone for Pediatric Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Madelyn Garcia, MD, MPH, University of Rochester, Dept of Emergency Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RSRB9986
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2008-07

CONDITIONS: Appendicitis; Child; Contrast Media
Keywords: Appendicitis; Computed tomography; pediatric; child; sensitivity; specificity; contrast administration route; time factors
MeSH Terms: conditions — Appendicitis; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): cohort = pediatric patients in the ED (3-18 yo) with abdominal pain suspicious for appendicitis that are to undergo CT scan
  Interventions: Other: CT Scan using IV contrast alone

INTERVENTIONS:
Other: CT Scan using IV contrast alone — CT scan using IV contrast alone

SUMMARY:
Computed tomography (CT) scan using intravenous contrast (CT IV) as the sole type of contrast material, was studied as one method of evaluating children with suspected appendicitis. We felt that this technique could provide physicians with a faster and better-tolerated alternative to CT imaging which involves patients drinking oral contrast or needing rectal contrast administered.

SPECIFIC AIMS

1. To test an imaging protocol using CT IV for the evaluation of suspected appendicitis in children in the setting of a pediatric emergency department (ED).
2. To determine test performance characteristics (specificity, sensitivity and diagnostic accuracy) of CT IV in detecting appendicitis in children.

DETAILED DESCRIPTION:
This was to be a prospective cohort study imaging pediatric patients (3-18 years old) in whom the diagnosis of appendicitis was suspected, but not clinically apparent. Patients that were to have a CT performed would be invited to participate and if enrolled, would be imaged using CT scan with IV contrast alone.

CT scans would be interpreted in real time by a resident radiologist and/or an attending radiologist. ED evaluation would remain unchanged and patient disposition would be based on the discretion of the ED provider using all information (patient exam, labs, surgical consultation as needed and the results of the CT scan).

CT scan performance would be determined by comparison of the CT interpretation with patient final outcomes as determined by either (1) pathology reports - in patients that went on to have surgery (appendectomy) or (2) clinical phone follow up at 24 hrs and then 1 week after ED discharge.

Performance of CT would be compared between the resident and the attending radiologists.

Further, we would compare the time to obtain a CT scan (defined as ED triage time - Time to CT) between our study cohort and a retrospective cohort of patients who had received CT scan in the ED for evaluation of appendicitis pre-study (CT using BOTH IV and oral contrast).

ELIGIBILITY:
Inclusion Criteria:

* Age 3- 18 years
* Signs/symptoms for < 72 hours
* CT Scan requested for evaluation by attending or fellow

Exclusion Criteria:

* Clinically apparent appendicitis
* Pregnancy
* Sickle Cell Disease
* Known contrast allergy
* Previous enrollment
* Signs/symptoms for > 72 hrs
* Known abdominal disease (e.g. Crohn's)
* Exam unreliable (neurologically impaired patient)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Actual)
Dates: Start 2003-11; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity, Specificity, PPV, NPV for CT Scan with IV contrast alone | Study completion date

SECONDARY OUTCOMES:
Time to CT scan for CT with IV contrast alone v. CT using both IV and oral contrast | study completion date

CONTACTS AND LOCATIONS:
Overall Officials: Madelyn Garcia, MD, MPH, Principal Investigator — University of Rochester; Lynn Babcock-Cimpello, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States